CLINICAL TRIAL: NCT07371182
Title: A Multi-center, Open-label, Single-arm Study of Luvometinib Monotherapy in Pediatric Langerhans Cell Histiocytosis With Single-system Special-site Single and Multifocal Bone Involvement
Brief Title: Luvometinib in Pediatric SS-LCH With Special-site Single/Multifocal Bone Lesions
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: West China Second University Hospital (Other)
Responsible Party: Principal Investigator, Ju Gao, Professor of Pediatrics, West China Second University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WCSH-NCP-SS-LCH-2026
Record Dates: First submitted 2026-01-18; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Langerhans Cell Histiocytosis (LCH)
MeSH Terms: conditions — Histiocytosis, Langerhans-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Luvometinib (Experimental)
  Interventions: Drug: Luvometinib

INTERVENTIONS:
Drug: Luvometinib — 5 mg/m² orally once daily for 1 year

SUMMARY:
Langerhans cell histiocytosis (LCH) is the most common type of histiocytic disorder in children, affecting about 2.6 to 8.9 out of every million kids each year. It can look very different from one child to another-some cases get better on their own-but when it affects special bones (like the base of the skull, temporal bone, eye socket, or spine) or when there are multiple bone lesions in one system, children often face a higher risk of long-term complications and the disease coming back.Current guidelines in China and around the world recommend treating these children with whole-body therapy, usually a chemotherapy combination of vinblastine and prednisone. However, even with longer treatment courses, about 27.6% of children with multiple bone lesions still have the disease return, and less than 70% stay free of events after 5 years. Some even develop lasting nerve system problems.

In recent years, researchers discovered that nearly all children with LCH have overactive MAPK signaling pathways in their cells. This discovery opened the door to using MAPK inhibitors as a new treatment. Studies have shown that these drugs work well and are safe for children with relapsed or hard-to-treat LCH. Even better, in some kids with single-system bone disease, the disease did not come back after stopping the drug-suggesting it might even cure certain cases.

Luvometinib (also called FCN-159), a new MAPK inhibitor developed by Fosun Pharma in Shanghai, was approved in 2025 for treating adult LCH. A Phase II clinical study showed very encouraging results: 82.8% of patients saw their disease improve or disappear, and 74.4% stayed free of progression after 12 months. The drug was well tolerated, with side effects that were mild and manageable-no serious problems forced anyone to stop treatment.Compared to traditional chemotherapy, luvometinib has fewer and milder side effects, does not weaken the immune system, and lets children continue normal daily life and school. It is a simple oral pill taken once a day, so there's no need for intravenous lines or hospital stays, making treatment much easier and improving quality of life for both the child and the family.

ELIGIBILITY:
Inclusion Criteria:

1. Children aged 0-18 years, both sexes.
2. Pathologically confirmed diagnosis of LCH (CD1a+ and/or CD207+), with no prior treatment specific to LCH.
3. Patients assessed as having single-system multifocal bone involvement, single-site bone involvement at central nervous system risk sites (central nervous system risk sites include craniofacial region [excluding parietal, occipital, and frontal bones], orbital, ear, and oral regions), or single-site vertebral bone involvement with intraspinal space-occupying lesion compressing the spinal cord.
4. Signed informed consent, willing to receive treatment according to this protocol and undergo follow-up.

Exclusion Criteria:

1. Patients with other underlying diseases, such as primary immunodeficiency, heart failure, renal insufficiency, hepatitis virus infection, HIV infection, post-organ transplantation, etc.
2. Secondary malignancy.
3. QTcF > 0.47 seconds on electrocardiogram prior to enrollment.
4. Ophthalmologic screening prior to enrollment reveals retinal vein occlusion, retinal pigment epithelial detachment, or other ocular diseases.
5. Patients with LCH carrying category 3 MEK mutations, specifically the following mutation sites: L98_I103del, L98_K104del, P105_A106del, P105_I107delinsL, L101_I103delinsF, E102_I103delinsF, E102_I103del, E102_I103delinsV, E102_I103delinsVN, E102_K104delinsQ, I103_A106del.
6. Refusal to sign the informed consent form.

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 62 (Estimated)
Dates: Start 2026-06-19 (Estimated); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Event-free survival rate | 2-year

SECONDARY OUTCOMES:
Objective response rate | 1 month and 3 month
Overall survival rate | 2-year
Safety of luvometinib | 1-year
Quality of life assessment in children | Before therapy，1month，3months，6months， 12months
Survey on satisfaction with drug treatment in children | Before therapy，1month，3months，6months， 12months

CONTACTS AND LOCATIONS:
Locations (11):
- China (11):
  - The Second Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - The Second Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - Affiliated Hospital of Guizhou Medical University, Guiyang, Guizhou
  - Zunyi Medical University Affiliated Hospital, Guizhou Provincial Children's Hospital, Zunyi, Guizhou
  - Jiangxi Provincial Children's Hospital, Nanchang, Jiangxi
  - Xi'an Children's Hospital, Xi'an, Shaanxi
  - Xi'an Northwest Women's and Children's Hospital, Xi'an, Shaanxi
  - West China Second Hospital, Sichuan University, Chengdu, Sichuan
  - The First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - Kunming Children's Hospital, Kunming, Yunan
  - Anhui Provincial Children's Hospital, Hefei

IPD SHARING:
Plan to Share IPD: No
IPD might be shared in the future upon approval by the ethics committee and under a data use agreement.

REFERENCES:
- [Result] Diamond EL, Emile JF, Fujino T, Haroche J, Maron MI, Lewis AM, Rahman J, Reiner AS, Bossert D, Rosenblum M, Yabe M, Petrova-Drus K, Francis JH, Rotemberg V, Rampal RK, Yoo S, Daniyan AF, Mahajan S, Hatzoglou V, Young R, Ulaner GA, Rosler W, Hershkovitz-Rokah O, Shpilberg O, Mazor RD, Chen LYC, Singer M, Cuibus MA, Weis K, Benbarche S, Zhang P, Fox N, Castro C, Tittley S, Witkowski M, Cohen-Aubart F, Terriou L, Hanoun M, Schleinitz N, Sosa G, Hautala T, De Lassus LF, Rosen N, Abdel-Wahab O, Durham BH. RAF-independent MEK mutations drive refractory histiocytic neoplasms but respond to ERK inhibition. Cancer Cell. 2026 Jan 12;44(1):203-220.e8. doi: 10.1016/j.ccell.2025.09.014. Epub 2025 Oct 23. PMID 41135521
- [Result] Cao XX, Zhu Q, Cai Z, Ma J, Zhou H, Chang L, Zhong LP, Wu ZL, Wang X, Han P, Lin HM, Wei Z, Guo JY, Zheng Y, Li J. Luvometinib in patients with Langerhans cell histiocytosis, Erdheim-Chester disease, and other histiocytic neoplasms: a single-arm, multicentre, phase 2 study. EClinicalMedicine. 2025 Sep 17;88:103486. doi: 10.1016/j.eclinm.2025.103486. eCollection 2025 Oct. PMID 41035796
- [Result] Keam SJ. Luvometinib: First Approval. Drugs. 2025 Sep;85(9):1177-1183. doi: 10.1007/s40265-025-02217-6. Epub 2025 Aug 2. PMID 40751881
- [Result] Whitlock JA, Geoerger B, Dunkel IJ, Roughton M, Choi J, Osterloh L, Russo M, Hargrave D. Dabrafenib, alone or in combination with trametinib, in BRAF V600-mutated pediatric Langerhans cell histiocytosis. Blood Adv. 2023 Aug 8;7(15):3806-3815. doi: 10.1182/bloodadvances.2022008414. PMID 36884302
- [Result] Cournoyer E, Ferrell J, Sharp S, Ray A, Jordan M, Dandoy C, Grimley M, Roy S, Lorsbach R, Merrow AC, Nelson A, Bartlett A, Picarsic J, Kumar A. Dabrafenib and trametinib in Langerhans cell histiocytosis and other histiocytic disorders. Haematologica. 2024 Apr 1;109(4):1137-1148. doi: 10.3324/haematol.2023.283295. PMID 37731389
- [Result] Donadieu J, Larabi IA, Tardieu M, Visser J, Hutter C, Sieni E, Kabbara N, Barkaoui M, Miron J, Chalard F, Milne P, Haroche J, Cohen F, Helias-Rodzewicz Z, Simon N, Jehanne M, Kolenova A, Pagnier A, Aladjidi N, Schneider P, Plat G, Lutun A, Sonntagbauer A, Lehrnbecher T, Ferster A, Efremova V, Ahlmann M, Blanc L, Nicholson J, Lambilliote A, Boudiaf H, Lissat A, Svojgr K, Bernard F, Elitzur S, Golan M, Evseev D, Maschan M, Idbaih A, Slater O, Minkov M, Taly V, Collin M, Alvarez JC, Emile JF, Heritier S. Vemurafenib for Refractory Multisystem Langerhans Cell Histiocytosis in Children: An International Observational Study. J Clin Oncol. 2019 Nov 1;37(31):2857-2865. doi: 10.1200/JCO.19.00456. Epub 2019 Sep 12. PMID 31513482
- [Result] Su M, Gao YJ, Pan C, Chen J, Tang JY. Outcome of children with Langerhans cell histiocytosis and single-system involvement: A retrospective study at a single center in Shanghai, China. Pediatr Hematol Oncol. 2018 Oct-Nov;35(7-8):385-392. doi: 10.1080/08880018.2018.1545814. Epub 2019 Jan 29. PMID 30693828
- [Result] Morimoto A, Shioda Y, Imamura T, Kudo K, Kitoh T, Kawaguchi H, Goto H, Kosaka Y, Tsunematsu Y, Imashuku S; Japan LCH Study Group. Intensification of induction therapy and prolongation of maintenance therapy did not improve the outcome of pediatric Langerhans cell histiocytosis with single-system multifocal bone lesions: results of the Japan Langerhans Cell Histiocytosis Study Group-02 Protocol Study. Int J Hematol. 2018 Aug;108(2):192-198. doi: 10.1007/s12185-018-2444-0. Epub 2018 Mar 28. PMID 29594922
- [Result] Haupt R, Minkov M, Astigarraga I, Schafer E, Nanduri V, Jubran R, Egeler RM, Janka G, Micic D, Rodriguez-Galindo C, Van Gool S, Visser J, Weitzman S, Donadieu J; Euro Histio Network. Langerhans cell histiocytosis (LCH): guidelines for diagnosis, clinical work-up, and treatment for patients till the age of 18 years. Pediatr Blood Cancer. 2013 Feb;60(2):175-84. doi: 10.1002/pbc.24367. Epub 2012 Oct 25. PMID 23109216
- [Result] Lin H, Batajoo A, Peckham-Gregory E, Zinn D, Eckstein OS, El-Mallawany NK, Gulati N, Prudowsky ZD, Scull B, Velazquez J, Abhyankar H, Simko SJ, Vakula D, Fleischmann R, Karri V, Hicks MJ, Fisher KE, Curry CV, Roy A, Schiff D, Heym KM, Scheurer ME, Parsons DW, Merad M, Man TK, McClain KL, Picarsic J, Allen CE. BRAF V600E-positive mononuclear cells in blood at diagnosis portend treatment failure and neurodegeneration in pediatric LCH. Blood. 2025 Jul 10;146(2):206-218. doi: 10.1182/blood.2024026671. PMID 40167581
- [Result] Rodriguez-Galindo C, Allen CE. Langerhans cell histiocytosis. Blood. 2020 Apr 16;135(16):1319-1331. doi: 10.1182/blood.2019000934. PMID 32106306